CLINICAL TRIAL: NCT06109337
Title: Immunoprofilling of Peripheral Blood Mononuclear Cells in Children With Attention Deficit/Hyperactivity Disorder
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstZhejiangU-fgh01
Record Dates: First submitted 2023-10-22; First posted 2023-10-31 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: ADHD; Immune System; Clinical Syndrome
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood monocyte
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD children: Take peripheral blood 5ml; IQ and cognitive function test; Head MRI scan
  Interventions: Diagnostic Test: drow blood
- typically developing controls: Take peripheral blood 5ml; IQ and cognitive function test; Head MRI scan
  Interventions: Diagnostic Test: drow blood

INTERVENTIONS:
Diagnostic Test: drow blood — Participants will be taken peripheral blood about 5 ml

SUMMARY:
The goal of this observational study is to learn about The immune cell landscape of peripheral blood mononuclear cells in children with ADHD compared to typically developing controls. The main question it aims to answer are: 1.Testing the differences in immune cell subpopulations, protein expression and signaling pathways and cell subsets between two groups 2. Exploring the correlations between immune function in PBMC and resting-state brain functional networks in children with ADHD.

Participants will be taken peripheral blood about 5 ml , cognitive assessment including Intelligence testing, Stroop color-word test and Trail making test, clinical interview and brain structural and functional MRI.

DETAILED DESCRIPTION:
3.1 Research Content Peripheral blood mononuclear cells of ADHD children and control group were taken, and 41 protein Marker on the cell surface was detected and analyzed by mass spectrometry flow cytometry (CyTOF) technology to draw a detailed map of ADHD immune cells, so as to explore the differences in protein expression level and subgroup distribution of immune cells between ADHD children and normal children. To evaluate the clinical symptoms, cognitive function, head MRI structure and resting state data of children with ADHD, and explore the correlation between immunophenotype and symptom score, cognition and brain structure.

3.2 Research Scheme 3.2.1 Collection of general and demographic data Demographic and clinical data, including name, age, sex, height, weight, age of first onset, course of disease, treatment, family history, past history and personal history, were collected by self-designed general situation scale.

3.2.2 Clinical evaluation The primary Clinical diagnosis was made by child psychiatrists with the title of attending psychiatrist or above through non-prescriptive clinical Interview, and the Clinical Diagnostic Interview Scale prepared by the American Working Group on Childhood Disorders was used. CDIS were conducted to evaluate ADHD classification, comorbidities, classification, comorbidities and clinical symptoms.

3.2.3 Core symptoms of ADHD ADHD-RS symptom assessment questionnaire was used to assess the severity of symptoms. The sum of scores of items in the attention deficit dimension is the attention deficit score, the sum of scores of items in the hyperactivity and impulsivity dimension is the score of hyperactivity impulse, and the sum of scores of all items is the score of the full scale. The higher the score, the more severe the symptoms.

3.2.4 Wechsler Intelligence test The Chinese children's Intelligence Scale (the third edition) was used to assess the IQ of the children.

3.2.5 Stroop color word naming test The test is divided into four parts. Part 1 asked the subjects to read red yellow green blue black character 6 Part 2 asked to name 30 red yellow green blue block colors; The third part requires reading 30 words whose meaning is inconsistent with the color of the print; Part 4 requires 30 read colors for word meaning and print color inconsistencies. The calculation indicators are: the completion time and the number of errors for each part. The results of part 1 and 2 reflect the ability of immediate attention; The time of Part 3 subtracts the time of Part 1 when the color interferes; The time of Part 4 minus the time of Part 2 is when the word is disturbed.

3.2.6 Trail making test (TMT) It is divided into A and B. In Formula A, the subjects were presented with numbers ranging from 1 to 25 randomly distributed, and were asked to connect the numbers accurately and quickly in an increasing order of 1-2-3 digits. The calculation measures the time and number of errors of the operation: reflects the visual spatial scanning and writing ability. In Formula B, the numbers 1-13 and letters A-L were distributed randomly and irregularly, and the subjects were required to accurately and quickly connect the numbers and letters in the cross order of 1-A-2-B-3-C. The calculation index was operation time and number of errors: the speed of reaction operation and the quality of completion. Use time B - time A: The ability to reflect the conversion of the subject.

3.2.7 The brain MRI structure and resting state data of subjects were collected High-resolution brain structure images were obtained using the Magnetization Prepared Rapid Acquisition Gradient-echo (MPRAGE) sequence with the following parameters: TR/TE= 7.1/2.9ms; sli-ces=146; Thickness =1 mm; Turnover Angle =8°; Matrix =256×256; Field of view =260×260 mm2; Voxel size 1*1*1mm.

Fmri images were collected by spin-echo-echo planar imaging (SE-EPI). The specific parameters were as follows: TR/TE=1800/30ms, section =28, thickness =4mm; Matrix =64×64, FOV=240×240 mm2, gap =0.8mm; Time point =180.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ADHD； Children with an IQ≥70； Both parents are Han； Agree to take venous blood with informed consent；

Exclusion Criteria:

Schizophrenia, mood disorder, autism, mental retardation； Obvious physical and nervous system abnormalities；

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and teenagers ages 6-12 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the differences in immune cell subpopulations, protein expression , signaling pathways between ADHD and typically developing children | 2023.11.1-2023.12.31 Participant recruitment and deta collections
  Blood samples of ADHD patients and normal control groups were collected, peripheral blood mononuclear cells were extracted, and 41 protein markers on cell surface were detected and analyzed by CyTOF technology, and detailed atlas of ADHD immune cells were drawn for immunological index analysis. These indicators include cytokine levels, immune cell subsets, and immune-related gene expression.
Clinical assessment and cognitive function testing | 2023.11.1-2023.12.31 Participant recruitment and deta collections
  The Clinical Diagnostic Interview Scale (CDIS) was used to evaluate ADHD types, comorbidities, types, comorbidities and clinical symptoms by child psychiatrists with the title of attending psychiatrist or above. ADHD-RS symptom assessment questionnaire was used to assess the severity of symptoms. Cognitive function tests include child IQ, Stroop color word naming test, and Trail making test (TMT).
Brain MRI structure and resting state data | 2023.11.1-2023.12.31 Participant recruitment and deta collections
  High-resolution brain structure images were acquired using 3D Magnetization Prepared Rapid Acquisition Gradient-echo (MPRAGE).
  The FMRI images were acquired by spin-echo-echo planar imaging (SE-EPI)

SECONDARY OUTCOMES:
General and demographic data collection | 2023.11.1-2023.12.31 data collection
  A comprehensive questionnaire included name, age, sex, height, weight, age of first onset, course of disease, treatment, family history, past history, personal history

CONTACTS AND LOCATIONS:
Overall Officials: Hu Guanghui, doctor, Principal Investigator — Department of Psychiatry, the First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Fu Guanghui, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ni Chasaide C, Lynch MA. The role of the immune system in driving neuroinflammation. Brain Neurosci Adv. 2020 Jan 29;4:2398212819901082. doi: 10.1177/2398212819901082. eCollection 2020 Jan-Dec. PMID 32219178
- [Result] Darwish AH, Elgohary TM, Nosair NA. Serum Interleukin-6 Level in Children With Attention-Deficit Hyperactivity Disorder (ADHD). J Child Neurol. 2019 Feb;34(2):61-67. doi: 10.1177/0883073818809831. Epub 2018 Nov 15. PMID 30430896